CLINICAL TRIAL: NCT03329898
Title: Randomized, Controlled Trial to Assess the Efficacy of Disposable Balloon Uterine Stent Combined With Estrogen or Dried Biological Amnion Graft in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Brief Title: Comparing the Efficacy of Two Methods for the Therapy of Uterine Adhesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: No.4-20171020
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Intrauterine Adhesion
Keywords: Asherman syndrome; uterine stent; hysteroscopy
MeSH Terms: conditions — Gynatresia | interventions — Estradiol; Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dried biological amnion graft (Experimental): dried biological amnion graft patients, who are with IUA, treated by uterine application of dried biological amnion graft + disposable balloon uterine stent + hormones (estradiol valerate tablets+dydrogesterone Tablets) following hysteroscopic adhesiolysis.
  Interventions: Procedure: dried biological amnion graft; Device: disposable balloon uterine stent; Drug: estradiol valerate tablets; Drug: dydrogesterone Tablets
- disposable balloon uterine stent only (Sham Comparator): disposable balloon uterine stent patients, who are with IUA, treated by uterine application of disposable balloon uterine stent only + hormones (estradiol valerate tablets+dydrogesterone Tablets) following hysteroscopic adhesiolysis.
  Interventions: Device: disposable balloon uterine stent; Drug: estradiol valerate tablets; Drug: dydrogesterone Tablets

INTERVENTIONS:
Procedure: dried biological amnion graft — dried biological amnion graft. The amnion grafts were spread on the balloon end of disposable balloon uterine stent .
  Other Names: uterine application of amnion membrance
  Arms: dried biological amnion graft
Device: disposable balloon uterine stent — the disposable balloon uterine stent is heart-shaped that resembled the shape of the uterine cavity and could fully separate the two sides of the uterine wall and the corners of the uterus.
Drug: estradiol valerate tablets — oral estradiol valerate tablets, which can promote endometrial growth after operation.
  Other Names: Progynova
Drug: dydrogesterone Tablets — oral dydrogesterone Tablets
  Other Names: Duphaston

SUMMARY:
Asherman's syndrome is characterized by the presence of intrauterine adhesions (IUA) as well as symptoms such as amenorrhea, hypomenorrhea, pelvic pain, and infertility. The gold standard for the treatment of intrauterine adhesions is hysteroscopic intrauterine adhesions. The recurrence of intrauterine adhesions is a major challenge in clinical practice. It has been reported that dried biological aminion graft was used to prevent adhesion after the operation of intrauterine adhesions. Intrauterine balloon can reduce the recurrence of adhesions after operation. Does the combination of balloon and amniotic products can improve clinical outcomes? Therefore, this study was conducted.

DETAILED DESCRIPTION:
The diaposable balloon uterine(a special intrauterine balloon) is usually inserted into the uterine after a hysteroscopic adhesiolysis and removed after on the 7th day after surgery. Another group, the diaposable balloon uterin and dried biological amnion will be inserted into the uterine after a hysteroscopic adhesiolysis and removed after on the 7th day after surgery.Several investigators demonstrated its favorable effect in the recurrence of adhesion after the treatment of intrauterine adhesion. Disposable balloon uterine stent is specially designed to fit into the cavity of the uterus, and usually removed on the 7th day after surgery.

Allocation: Randomized Endpoint Classification: Safety/Efficacy Study Intervention Model: Parallel Assignment Masking: Single Blind (Subject) Primary Purpose: Prevention

ELIGIBILITY:
Inclusion Criteria:

* age 20-45 years.
* previously diagnostic hysteroscopy confirmed adhesion score ≧5， according to the American Fertility Society (AFS).
* complains of menstruation disorder and reproductive dysfunction.
* informed consent.

Exclusion Criteria:

* premature menopause,
* presence of other intrauterine lesions (e.g. polyps, myoma, septa), and
* presence of severe intercurrent illness (e.g. systemic disease, coagulative disorders, severe kidney and liver diseases),
* adhesions limited to the lower uterine cavity or the cervical canal.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-10-25 (Estimated); Study Completion 2018-11-25 (Estimated)

PRIMARY OUTCOMES:
second diagnostic hysteroscopy | postoperation three months
  American fertility society score ,Scores of 1-4, 5-8, and 9-12 were considered to represent mild, moderate, and severe adhesions, respectively

SECONDARY OUTCOMES:
pregnancy | postoperation one year
  the number of biochemical pregnancy or clinical pregnancy
Menstruation Pattern | postoperation three months
  Amenorrhoea, hypomenorrhea, normal menstrual volume
adhesion reformation | postoperation three months
  Adhesion is seen under direct vision by hysteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Duan Hua, PhD, Study Chair — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided